CLINICAL TRIAL: NCT03040011
Title: Preoperative Levator Ani Muscle Injection and Pudendal Nerve Block With Bupivacaine and Dexamethasone for Improved Pain Control After Vaginal Reconstructive Surgery: A Three-Arm Randomized Controlled Trial
Brief Title: Preoperative Levator Ani Muscle Injection and Pudendal Nerve Block for Pain Control After Vaginal Reconstructive Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lauren Giugale, MD (Other)
Collaborators: Magee-Women's Research Institute (Other)
Responsible Party: Sponsor-Investigator, Lauren Giugale, MD, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO16110378
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Organ Prolapse; Surgery; Postoperative Pain
Keywords: Vaginal Surgery; Pelvic Organ Prolapse; Postoperative Pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain, Postoperative | interventions — Dexamethasone; Calcium Dobesilate; Bupivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Three-arm, double-blinded, placebo-controlled, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupivacaine/Dexamethasone Arm (Experimental): After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen (transobturator). After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of a mixture of 20 milliliters of 0.25% bupivacaine (2.5mg/milliliter ) and 2 milliliters of dexamethasone (4mg/milliliter). The total amount of the bupivacaine/dexamethasone solution will be divided equally between the four injection sites.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Procedure: Bilateral Pudendal Nerve Block; Procedure: Bilateral Levator Ani Muscle Injection
- Bupivacaine Arm (Active Comparator): After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen (transobturator). After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of 20 milliliters 0.25% bupivacaine (2.5mg/milliliter). The total amount will be divided equally between the four injection sites.
  Interventions: Drug: Bupivacaine; Procedure: Bilateral Pudendal Nerve Block; Procedure: Bilateral Levator Ani Muscle Injection
- Placebo Arm (Placebo Comparator): After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen (transobturator). After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of 20 milliliters 0.9% saline (normal saline). The total amount will be divided equally between the four injection sites.
  Interventions: Procedure: Bilateral Pudendal Nerve Block; Procedure: Bilateral Levator Ani Muscle Injection; Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Other Names: Decadron
  Arms: Bupivacaine/Dexamethasone Arm
Drug: Bupivacaine — Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Other Names: Marcaine
  Arms: Bupivacaine Arm; Bupivacaine/Dexamethasone Arm
Procedure: Bilateral Pudendal Nerve Block — Performed transvaginally. The ischial spines will be palpated transvaginally and the sacrospinous ligament identified as a firm band running medially and posteriorly from the ischial spine to the sacrum. The needle guide will be inserted and positioned against the vaginal mucosa on the sacrospinous ligament approximately 1 cm medial and inferior to the ischial spine. When the needle guide is properly positioned, the spinal needle is advanced approximately 1cm through the vaginal mucosa into the sacrospinous ligament. The needle will be aspirated to ensure no intravascular needle placement. With a negative aspirate, 5 milliliters of solution are injected. This same procedure will be performed on the contralateral side.
Procedure: Bilateral Levator Ani Muscle Injection — Performed transperineally. With thumb, superomedial aspect of obturator foramen is palpated 2-3 cm lateral to the clitoris. The index and middle finger are in the vagina to confirm obturator foramen. A spinal needle is inserted through the the obturator foramen into the obturator internus muscle. The needle is angled slightly posteriorly towards the ischial spine, parallel to the arcus tendineus levator ani and arcus tendineus fascia pelvis. The needle is advanced to the level of the ischial spine, the vaginal hand ensuring that the needle has not perforated the vaginal wall. Once the needle tip is at a depth of the ischial spine, aspiration is performed to ensure no intravascular needle placement. 5 milliliters of solution is injected along the length of the needle tract.
Drug: Saline — Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Other Names: Normal Saline
  Arms: Placebo Arm

SUMMARY:
To test the hypothesis that preoperative injections along the levator ani muscles and pudendal nerve with bupivacaine and dexamethasone improve pain control after vaginal apical reconstructive surgery. A three-arm, double-blinded, randomized controlled trial of a total of 75 women will be performed.

The study population will be adult women (>18 years of age) with uterovaginal or vaginal vault prolapse who have been scheduled for native tissue vaginal reconstructive surgery which includes an apical support procedure. Participants will be enrolled prior to surgery. The procedure will involved four injection sites: the bilateral levator ani muscles via a transobturator approach and bilateral pudendal nerves via a transvaginal approach. Random assignment will occur to one of three study arms: combined arm (20 milliliters bupivacaine/dexamethasone solution divided between the 4 injection sites), bupivacaine arm (20 milliliters bupivacaine divided between the 4 injection sites), or placebo arm (20 milliliters saline divided between the 4 injection sites).

DETAILED DESCRIPTION:
The primary purpose of this three arm, randomized clinical trial is to test the hypothesis that preoperative injections along the levator ani muscles and pudendal nerve with bupivacaine and dexamethasone improve pain control after vaginal native tissue apical reconstructive surgery.

Hypothesis: concurrent bilateral transobturator levator ani muscle injections and transvaginal pudendal nerve blocks with bupivacaine and dexamethasone performed prior to vaginal apical support procedures will result in improved pain scores at 24 hours postoperatively.

Participants will be randomized to three arms: bupivacaine/dexamethasone group, bupivacaine group, and placebo group. Block randomization will occur and will be stratified by surgery type to ensure that similar numbers of each procedure are randomized to each study arm.

All 3 groups will receive pudendal nerve blocks and transobturator levator ani muscle injections as outlined in detail below (with either bupivacaine/dexamethasone, bupivacaine alone or saline depending on randomization). The interventions will be performed after the participant is positioned in lithotomy position and after sterile preparation of the vagina and perineum per standard protocol. These injections will be performed at the start of the procedure prior to any vaginal repair and be administered by either the attending surgeon or the urogynecology fellow. After the interventions below, the vaginal reconstructive procedures will be performed as usual by the attending surgeon and surgical team. There are both fellows and residents who participate in these vaginal reconstructive surgeries, however for study purposes, resident physicians will not be permitted to administer either the pudendal nerve block or the transobturator injections. There are four attending surgeons and four fellow physicians who will be administering the injections. While all surgeons are familiar with the anatomy and have performed these procedures, each physician will be instructed on the intended procedures and additionally will be directly observed in the operating room for at least one procedure to ensure consistency in technique. All participants will undergo a standardized general anesthesia regimen.

After the study intervention, all participants will then undergo the scheduled vaginal reconstructive procedure as standard. Infiltration of the vaginal epithelium with lidocaine is common in vaginal repairs. The maximum doses of lidocaine and bupivacaine are additive. The amount of local infiltration to 50 milliliters of 0.5% lidocaine with epinephrine. This dose is equal to 250mg of lidocaine which, when also taking into account the 50mg of bupivacaine, is within a safe dosing range for a participant weighing 50kg.

Administration of all four injections involved in the study protocol and described above take approximately 5 additional minutes in total at the start of the case. After the injections are performed, there will be no further interventions.

Other assessments that will be performed as part of the study protocol are outlined below:

Baseline assessments: Pain assessment, assessment of presence of any baseline nausea or vomiting, baseline activities assessment will all be performed in preoperative area on the day of surgery prior to randomization.

Postoperative pain score assessment: 3 hours, 24 hours, 48 hours, 72 hours, and 1 week postoperatively. Postoperative pain measured by the numerical rating scale (NRS). The NRS is a publicly available pain assessment tool that consists of an eleven point scale ranging from 0 to 10 (0 = no pain and 10 = worst possible pain) presented visually on a horizontal line. Participants are asked to report a number or mark on the scale. Previous studies have demonstrated its reliability, validity and ease of administration. The NRS was chosen because a systematic review article demonstrated higher compliance rates, better responsiveness and ease of use relative to visual analog scales. Additionally, the NRS has been shown to have strong validity and low error rates when used in an elderly (>60 years) postoperative patient population.

Postoperative nausea and vomiting assessment: 3 hours postoperatively The intensity of postoperative nausea and vomiting (PONV) using the PONV Intensity scale. The PONV scale is a four question assessment designed to measure clinically significant nausea and vomiting. It was initially validated in a general surgery population and has been validated in early postoperative gynecology patients. Clinically important nausea and vomiting is defined as a score greater than or equal to 50. This scale takes approximately 1 minute to complete and is publicly available. The amount of inpatient anti-emetic consumption will also be assessed. Any anti-emetic administered from surgery end time will be recorded as well as the dosage. Anti-emetic type and dosage will be recorded until the time of discharge.

Voiding status at time of foley catheter removal. All patients routinely have some assessment of voiding function prior to discharge. Whether each participant passed or failed a voiding trial after surgery will be recorded in the database. If a participant fails, the standard of care is do be discharged to home after learning self-catheterization or with a foley catheter. In the event that a participant fails a postoperative voiding trial, whether participants receive a foley catheter or were performing self-catheterization will be recorded. As this is a routine part of postoperative care, the research protocol will not interfere with the performance or outcomes of a voiding trial. Results will be documented, however no specific assessment tool will be used.

Time to resume normal activities measured by the activities assessment scale (AAS): 1 week, 2 weeks, 6 weeks and 12 weeks postoperatively The AAS was initially designed to assess functional activity in the perioperative period in the general surgery population. It has since been deemed a valid and reliable measure to assess postoperative activity level in a Female Pelvic Medicine and Reconstructive Surgery patient population. It has the ability to measure perioperative function and takes approximately 3-5 minutes to complete. It consists of a 13 item questionnaire assessing various types of physical activity and the degree of difficulty associated with each activity. The types of activities assessed fall into three subscales: sedentary activities (questions 1-4), ambulatory activities (questions 6-8), and work or exercise activities (questions 11-13). Respondents also have the option to indicate that these activities were not performed for another indication (this item is not scored). The time frame for all questions is the previous 24 hours. Given that many patients are instructed to avoid strenuous work or exercise activity in the postoperative period, the subscales of sedentary activities and ambulatory activities, which patients are encouraged to perform as tolerated in the postoperative period, will be of most interest.

Consumption of analgesic medications: during inpatient hospital stay and for first 72 hours postoperatively Narcotic consumption will be measured in morphine equivalents. The amount of narcotics will be obtained from the inpatient hospital record. All narcotics received from the surgery end time to the time of discharge will be included. Morphine equivalents will be calculated with online calculator available at http://www.agencymeddirectors.wa.gov/Calculator/DoseCalculator.htm. Similarly, the amount of NSAIDs will be obtained from the inpatient hospital record. All NSAIDs received from the surgery end time to the time of discharge will be included. To assess both the amount of narcotic and NSAID consumption after discharge, the participant will be provided with a diary form to record how many daily tablets of narcotic and NSAIDs are taken. This form will be completed from postoperative days 1-3.

For all forms, the participants will be instructed to mail the forms back to the office once completed (in a pre-address envelope provided as part of the study). Participants will also have the option of brining the forms in to the office at the time of a participant's postoperative visit.

Participants, physicians and any nursing personnel involved in patient care will remain masked until 12 weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18 or older who are scheduled for a vaginal native tissue repair with apical support procedure including uterosacral ligament suspension, sacrospinous ligament fixation, or colpectomy and colpocleisis with or without levator myorrhaphy
2. Concomitant procedures including hysterectomy, anterior and posterior colporrhaphies , perineorrhaphies and midurethral sling placements are acceptable and do not result in exclusion
3. Available for at least 12 weeks of follow-up
4. Able to undergoing general anesthesia

Exclusion Criteria:

1. Planned mesh-augmented apical support procedure (placement of synthetic midurethral sling is acceptable and not considered an exclusion criteria)
2. Planned mesh excision
3. Laparoscopic, robotic or abdominal surgery
4. Known adverse reaction or allergy to intervention medication
5. Evidence of fistula or known infection (vulvovaginal cellulitis, abscess, abdominopelvic infection, or systemic fungal infection)
6. Chronic pelvic pain as an active issue
7. Daily opiate consumption for any indication
8. History of pelvic radiation
9. Chronic steroid use
10. Diabetes mellitus
11. Known HIV/AIDS or immunosuppression secondary to transplant related medications
12. Planned surgery under regional anesthesia
13. Non-English speaking or inability to complete questionnaires
14. Bleeding disorders that would impair a patient's clotting ability
15. Weight less than 50kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Giugale, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dexamethasone (systemic): Drug information. UpToDate; 2016. Accessed November 9, 2016.
- [Background] Bupivacaine: Drug Information. UpToDate; 2016.
- [Background] Hsu D. Infiltration of local anesthetics. UpToDate. 2016. Accessed November 30, 2016.
- [Derived] Giugale LE, Baranski LA, Meyn LA, Schott NJ, Emerick TD, Moalli PA. Preoperative Pelvic Floor Injections With Bupivacaine and Dexamethasone for Pain Control After Vaginal Prolapse Repair: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):21-31. doi: 10.1097/AOG.0000000000004205. PMID 33278291

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment but before randomization, 4 patients withdrew from the study: surgical location changed (n=1), declined to participate (n=1), unsafe for general anesthesia (n=1), reported lidocaine allergy (n=1). Because they withdrew prior to randomization, we received permission to enroll an additional 4 patients to meet goal sample size of 75.
Groups:
- Bupivacaine/Dexamethasone Arm: After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen. After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of a mixture of 20 milliliters of 0.25% bupivacaine (2.5mg/milliliter ) and 2 milliliters of dexamethasone (4mg/milliliter). The total amount of the bupivacaine/dexamethasone solution will be divided equally between the four injection sites.
  Dexamethasone: Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Bupivacaine: Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Bilateral Pudendal Nerve Block: Performed transvaginally. The ischial spines will be palpated transvaginally and the sacrospinous ligam
- Bupivacaine Arm: After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen. After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of 20 milliliters 0.25% bupivacaine (2.5mg/milliliter). The total amount will be divided equally between the four injection sites.
  Bupivacaine: Pudendal Nerve and Levator Muscle Injection. See additional information in study arm description.
  Bilateral Pudendal Nerve Block: Performed transvaginally. The ischial spines will be palpated transvaginally and the sacrospinous ligament identified as a firm band running medially and posteriorly from the ischial spine to the sacrum. The needle guide will be inserted and positioned against the vaginal mucosa on the sacrospinous ligament approximately 1 cm m
- Placebo Arm: After sterile preparation in lithotomy position, investigators will perform bilateral levator ani muscle injection via the obturator foramen. After transobturator injections are performed on each side, bilateral pudendal nerve blocks will be performed transvaginally as described in the literature. The solution injected at all 4 of the above injections sites will consist of 20 milliliters 0.9% saline (normal saline). The total amount will be divided equally between the four injection sites.
  Bilateral Pudendal Nerve Block: Performed transvaginally. The ischial spines will be palpated transvaginally and the sacrospinous ligament identified as a firm band running medially and posteriorly from the ischial spine to the sacrum. The needle guide will be inserted and positioned against the vaginal mucosa on the sacrospinous ligament approximately 1 cm medial and inferior to the ischial spine. When the needle guide is properly positioned, the spinal needle is advanced approx
Period: Received Randomized Study Intervention
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0
Period: Primary Outcome Follow Up
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Started | 25 | 25 | 25
Completed (Outcome data are provided for all patients who underwent study intervention by intention to treat.) | 21 (Postoperative day one pain score not available for four patients) | 24 (Postoperative day one pain score not available for one patient) | 24 (Postoperative day one pain score not available for one patient)
Not Completed | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (13.6) | 68.0 (10.1) | 70.2 (9.2) | 69.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 75
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 0 | 6
  White | 22 | 21 | 24 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75
Baseline NRS Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — Pain measured by the numerical rating scale (NRS) prior to surgery. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
  units on a scale | 0 [0 to 0] | 0 [0 to 0.3] | 0 [0 to 0] | 0 [0 to 0]
Baseline NV Score [Median (Inter-Quartile Range); unit: units on a scale] — Any preoperative nausea and vomiting was assessed by administering the Postoperative Nausea and Vomiting Intensity Scale prior to surgery. The Postoperative Nausea and Vomiting Intensity Scale is a four-question assessment to measure clinically significant nausea and vomiting with a range from 0-7 with higher scores signifying more clinically significant nausea and vomiting. We chose to utilize this scale before and after surgery for consistency.
  units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Baseline AAS Score [Median (Inter-Quartile Range); unit: units on a scale] — The AAS is a 13-point scale on which patients rate their difficulty performing a range of activities from "No difficulty" to "Not able to do it." A final score ranging from 0-100 is transformed, with higher numbers reflecting less difficulty with activities.
  units on a scale | 94.6 [85.2 to 100] | 92.3 [70.6 to 100] | 95.5 [81.3 to 100] | 94.2 [79.4 to 100.0]
Prolapse Procedure [Count of Participants; unit: Participants]
  Uterosacral Ligament Suspension | 4 | 8 | 11 | 23
  Sacrospinous Ligament Fixation | 2 | 3 | 3 | 8
  Colpocleisis | 14 | 9 | 7 | 30
  Levator Myorrhaphy | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Primary Postoperative Pain Measured by the Numerical Rating Scale (NRS)
Description: Postoperative pain measured by the numerical rating scale (NRS) at 24 hours postoperatively. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
Time Frame: 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 21 | 24 | 24
score on a scale | 3.0 [1.0 to 5.0] | 4.0 [2.0 to 5.0] | 3.75 [2.0 to 6.5]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.39, Kruskal-Wallis

2. Secondary Outcome: 6 Hour Postoperative Pain Measured by the NRS
Description: Postoperative pain as measured by the NRS at 6 hours after surgery. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
  Of note, there is a typographical error in the protocol section and refers to this outcome as a NRS score at 3 hours postoperatively. The final IRB approved protocol is a 6 hour postoperative timepoint and this is the correct outcome reported here in the results section.
Time Frame: 6 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 1.0 [0.5 to 4.0] | 3.0 [2.0 to 4.0] | 1.75 [0.6 to 4.0]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.25, Kruskal-Wallis

3. Secondary Outcome: POD 2 Postoperative Pain Measured by the NRS
Description: Postoperative Pain Measured by the NRS 2 days after surgery. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
Time Frame: 2 days after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 3.0 [1.0 to 5.0] | 3.0 [2.0 to 4.0] | 4.0 [2.8 to 6.0]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.17, Kruskal-Wallis

4. Secondary Outcome: POD 3 Postoperative Pain Measured by the NRS
Description: Postoperative Pain Measured by the NRS 3 days after surgery. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
Time Frame: 3 days after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 3.0 [2.0 to 5.0] | 2.5 [2.0 to 3.3] | 3.5 [0.5 to 5.8]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.45, Kruskal-Wallis

5. Secondary Outcome: 1 Week Postoperative Pain Measured by the NRS
Description: Postoperative Pain Measured by the Numeric Rating Scale 1 week after surgery. The Numeric Rating Scale is an 11 point scale ranging from 0-10 with higher scores indicating worse pain.
Time Frame: 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 1.75 [1.0 to 2.75] | 2.0 [1.0 to 4.0] | 1.0 [0.0 to 3.5]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.54, Kruskal-Wallis

6. Secondary Outcome: Proportion of Patients With Same Day Discharge
Description: Same day discharge was defined as a patient being discharged on the same day as surgery and did not require an admission after surgery. The proportion of patients who were discharged on the day of surgery was compared between groups.
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 20 | 22 | 20
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.80, Chi-squared

7. Secondary Outcome: Postoperative Urinary Retention
Description: Urinary retention was defined as the need to perform self-catheterization or have an indwelling catheter placed postoperatively. The proportion of patients with urinary retention was compared between groups.
Time Frame: 0-24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 13 | 11 | 14
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.72, Chi-squared

8. Secondary Outcome: Adverse Events
Description: The number of adverse events in each study group was assessed and compared between study groups. An adverse event was described as any medical or surgical complication that occurred either intraoperatively or postoperatively.
Time Frame: 0-12 weeks postoperatively
Measure: Number; unit: number of adverse events
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
number of adverse events | 7 | 6 | 9
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.64, Chi-squared

9. Secondary Outcome: Nausea and Vomiting Measured by the PONV Scale
Description: Intensity of postoperative nausea and vomiting (PONV) measured by the PONV scale prior to discharge. The Postoperative Nausea and Vomiting Intensity Scale is a four-question assessment to measure clinically significant nausea and vomiting with a range from 0-7 with higher scores signifying more clinically significant nausea and vomiting.
Time Frame: 6 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.41, Kruskal-Wallis

10. Secondary Outcome: Anti-emetic Consumption
Description: The amount of inpatient anti-emetic consumption, recorded in number of doses of nausea medication
Time Frame: 3 hours postoperatively
Population: This data was not collected. Rather, we assessed the PONV score which is described in outcome number 9.
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Return to Baseline Activities Using the Activities Assessment Scale
Description: Resumed normal daily activities using the Activities Assessment Scale (AAS) by 1 week after surgery. The AAS is a 13-point scale on which patients rate their difficulty performing a range of activities from "No difficulty" to "Not able to do it." A final score ranging from 0-100 is transformed, with higher numbers reflecting less difficulty with activities.
  We defined return to normal as when a patient's postoperative AAS scores was at or greater than the baseline AAS score. We report the proportion of patients in each study arm who returned to baseline activity at each timepoint.
Time Frame: 1 week postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 11 | 11 | 12
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.96, Chi-squared

12. Secondary Outcome: Return to Baseline Activities Using the Activities Assessment Scale
Description: Resumed normal daily activities using the Activities Assessment Scale (AAS) by 2 weeks after surgery. The AAS is a 13-point scale on which patients rate their difficulty performing a range of activities from "No difficulty" to "Not able to do it." A final score ranging from 0-100 is transformed, with higher numbers reflecting less difficulty with activities.
  We defined return to normal as when a patient's postoperative AAS scores was at or greater than the baseline AAS score. We report the proportion of patients in each study arm who returned to baseline activity at each timepoint.
Time Frame: 2 week postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 15 | 16 | 14
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.90, Chi-squared

13. Secondary Outcome: Return to Baseline Activities Using the Activities Assessment Scale
Description: Resumed normal daily activities using the Activities Assessment Scale (AAS) by 6 weeks after surgery. The AAS is a 13-point scale on which patients rate their difficulty performing a range of activities from "No difficulty" to "Not able to do it." A final score ranging from 0-100 is transformed, with higher numbers reflecting less difficulty with activities.
  We defined return to normal as when a patient's postoperative AAS scores was at or greater than the baseline AAS score. We report the proportion of patients in each study arm who returned to baseline activity at each timepoint.
Time Frame: 6 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 19 | 17 | 17
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.49, Chi-squared

14. Secondary Outcome: Return to Baseline Activities Using the Activities Assessment Scale
Description: Resumed normal daily activities using the Activities Assessment Scale (AAS) by 12 weeks after surgery. The AAS is a 13-point scale on which patients rate their difficulty performing a range of activities from "No difficulty" to "Not able to do it." A final score ranging from 0-100 is transformed, with higher numbers reflecting less difficulty with activities.
  We defined return to normal as when a patient's postoperative AAS scores was at or greater than the baseline AAS score. We report the proportion of patients in each study arm who returned to baseline activity at each timepoint.
Time Frame: 12 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
Participants | 21 | 19 | 18
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.19, Chi-squared

15. Secondary Outcome: POD 1 Narcotic Consumption
Description: The total amount of narcotic pain medication used on postoperative day 1 was calculated and measured in oral morphine equivalents.
Time Frame: Postoperative day 1
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
oral morphine equivalents | 7.5 [0.0 to 15.0] | 4.4 [0.0 to 10.0] | 7.5 [0.0 to 22.5]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.35, Kruskal-Wallis

16. Secondary Outcome: POD 2 Narcotic Consumption
Description: The total amount of narcotic pain medication used on postoperative day 2 was calculated and measured in oral morphine equivalents.
Time Frame: Postoperative day 2
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
oral morphine equivalents | 7.5 [0.0 to 15.0] | 0.0 [0.0 to 11.9] | 7.5 [0.0 to 20.6]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.32, Kruskal-Wallis

17. Secondary Outcome: POD 3 Narcotic Consumption
Description: The total amount of narcotic pain medication used on postoperative day 3 was calculated and measured in oral morphine equivalents.
Time Frame: Postoperative day 3
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
oral morphine equivalents | 7.5 [0.0 to 15.0] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 18.8]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.18, Kruskal-Wallis

18. Secondary Outcome: POD 1 Ibuprofen Consumption
Description: The total amount of ibuprofen medication used on postoperative day 1.
Time Frame: Postoperative day 1
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
milligrams | 1200 [0 to 2400] | 1200 [750 to 1800] | 1200 [0 to 1800]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.68, Kruskal-Wallis

19. Secondary Outcome: POD 2 Ibuprofen Consumption
Description: The total amount of ibuprofen medication used on postoperative day 2.
Time Frame: Postoperative day 2
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
milligrams | 1200 [0 to 2400] | 1200 [750 to 1800] | 1800 [300 to 2400]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.40, Kruskal-Wallis

20. Secondary Outcome: POD 3 Ibuprofen Consumption
Description: The total amount of ibuprofen medication used on postoperative day 3.
Time Frame: Postoperative day 3
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 25 | 25 | 25
milligrams | 1200 [0 to 2400] | 1200 [0 to 2250] | 1800 [150 to 2400]
Statistical Analysis 1: Comparison: Bupivacaine/Dexamethasone Arm vs Bupivacaine Arm vs Placebo Arm; Test type: Superiority; p = 0.44, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 12 weeks from the date of surgery
Description: Members of the study team including the PI, research staff and coordinator met monthly. Any adverse event that was significant, unexpected and possibly related to the study procedure or medication was reported to the PI, faculty mentor and the IRB within 24 hours. The PI submitted in writing to the IRB a detailed summary of the adverse events for review. After IRB review of the adverse events, a final conclusion and recommendation were provided.
Arm/Group | Bupivacaine/Dexamethasone Arm | Bupivacaine Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 2/25
Other Adverse Events (participants affected / at risk) | 6/25 | 6/25 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine/Dexamethasone Arm (N=25) | Bupivacaine Arm (N=25) | Placebo Arm (N=25)
Surgical complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) — Surgical complications not thought to be related to study intervention: ureteral obstruction requiring return to the operating room (n=1) and a case with a rectal injury and sponge miscount, which was resolved prior to the procedure conclusion (n=1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Postoperative asthma exacerbation requiring emergency room care
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine/Dexamethasone Arm (N=25) | Bupivacaine Arm (N=25) | Placebo Arm (N=25)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) — Postoperative urinary tract infection defined as positive urine culture with symptoms
Excess postoperative surgical pain (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) — Excessive postoperative surgical site pain that required additional visits and medications
Intraoperative bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Bradycardia that required additional medication. Occurred after anesthesia but prior to the start of the surgical procedure. Not thought to be related to study intervention.
Leg numbness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) — Transient lower extremity numbness requiring extended observation and ultimately resolved spontaneously
Nausea and vomiting, diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — Postoperative nausea and vomiting and diarrhea on that required observation and medication administration. Not thought to be related to study intervention.
Fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Presented to emergency room with low grade fever of 100.4 Fahrenheit. Complete evaluation with no evidence of infection or other source of fever. No treatment or intervention required. Not thought to be related to study intervention.
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Fell at home one week after surgery requiring evaluation in emergency room. Not thought to be related to study intervention.
Yeast Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Vulvar yeast infection requiring medication. Not thought to be related to study intervention.
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Postoperative malodorous discharge and fever presumed wound infection (no culture obtained). Treated with antibiotics with symptom resolution. Not thought to be related to study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03040011/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT03040011/ICF_001.pdf